CLINICAL TRIAL: NCT00860457
Title: Lenalidomide Following Rituximab and Fludarabine in Untreated Chronic Lymphocytic Leukemia
Brief Title: Lenalidomide Following Fludarabine/Rituximab (FR) in Untreated Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-CLL-PI-089
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2014-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Rituximab; fludarabine; fludarabine phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Fludarabine/Rituximab followed by Lenalidomide
  Interventions: Drug: Rituximab; Drug: Fludarabine; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 IV infusion Day 1 of each 28-day cycle for maximum of 6 cycles
  Other Names: Rituxan
Drug: Fludarabine — 25 mg/m2 IV Days 1-5 of each 28-day cycle for maximum of 6 cycles
  Other Names: Fludara
Drug: Lenalidomide — 5-10 mg PO daily on Days 1-21 of each 28-day cycle for a maximum of 6 cycles
  Other Names: Revlimid

SUMMARY:
This study is for patients with chronic lymphocytic leukemia (CLL) who have not yet received any treatment for their disease.

Current therapy for this disease includes the use of combination chemotherapy regimens containing Fludarabine and Rituximab, which have been found to be very effective for CLL. In this study, subjects will receive Fludarabine and Rituximab. After 3 cycles or 6 cycles of Fludarabine and Rituximab treatment, they will receive Lenalidomide. We are doing this research because we are attempting to improve the response, or outcome, of Fludarabine and Rituximab in previously untreated CLL patients. Lenalidomide is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Lenalidomide is approved by the Food and Drug Administration (FDA) for treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM). MDS and MM are blood disorders that involve different types of blood cells. It is not approved for chronic lymphocytic leukemia. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental.

This research is being done because we are attempting to find a better treatment for chronic lymphocytic leukemia. We do not know the effect of Lenalidomide following the regimen of Fludarabine and Rituximab.

The hypothesis of the study is that adding Lenalidomide after the standard treatment regimen of Fludarabine and Rituximab will have better outcomes than treatment with Fludarabine and Rituximab alone.

DETAILED DESCRIPTION:
This is a single institution Phase II study where all enrolled patients with untreated CLL will receive fludarabine and rituximab (FR) combination therapy. Subjects who demonstrate Stable disease or Progressive disease after completing 3 cycles of FR will receive lenalidomide monotherapy for a maximum of 6 cycles. Subjects who achieve >/= PR after receiving 3 cycles of FR will receive 3 additional cycles of FR (maximum of 6 cycles). Upon completion of FR treatment subjects will receive lenalidomide monotherapy for a maximum of 6 cycles.

Response assessment will be performed for Module A (FR): after every cycle, but would include imaging after cycle 3 if clinically indicated. Response assessment will be performed for Module B (Lenalidomide monotherapy): Before starting Lenalidomide therapy, after every cycle and on completion of therapy. Imaging for Module B would be obtained before starting lenalidomide therapy, and on completion of therapy. Bone marrow biopsies will be performed prior to starting therapy in Module A (FR), prior to starting Module B (Lenalidomide), and on completion of Module B. Bone marrow biopsies can be obtained once during Lenalidomide therapy at the discretion of the investigator. Minimum residual disease assessment of bone marrow specimens should include immunohistochemistries and flow cytometry. Additional studies on bone marrow specimens will be sent for flow cytometric analysis (standard or four color flow), ZAP-70 immunohistochemical stains and FISH analysis (13q deletion, trisomy 12, 11q deletion, and 17p) will be performed at the time intervals described above.

Response will be assessed according to the Cheson Criteria.

Blood specimens for optional correlative studies will be drawn on Day 0 prior to FR, prior to starting lenalidomide, 90 days after initiation of lenalidomide, and 7 days after the last dose of lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign informed consent form
* No prior therapy for CLL
* Able to adhere to study visit schedule and other protocol requirements
* CLL with any Rai Stage requiring therapy
* ECOG performance status </= 2
* Absolute neutrophil count >/= 1.0
* Platelet count >/= 75
* Serum creatinine </= 1.5
* Total bilirubin </= 1.5
* AST and ALT </= 2 x ULN
* Females of childbearing potential must have negative pregnancy test
* Disease free of prior malignancies for >/= 5 years
* Able to take aspirin daily as prophylactic anticoagulation

Exclusion Criteria:

* Any serious medical condition, lab abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or lactating females
* Any condition, including the presence of lab abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV or infectious active hepatitis, type A, B
* Known hypersensitivity to nucleoside analogue or rituximab
* Previous treatment for CLL prior to enrolling in study
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Active hemolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Cheson, MD, Principal Investigator — Georgetown University
Locations (1):
- Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy
Started | 22
Completed | 11
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 60.5 [41 to 78]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Response assessments were made per the NCI working group criteria for CLL (Hallek et al, Blood, 2008). Complete response rate is defined as an achievement of all of the following: Peripheral blood lymphocytes (evaluated by blood and differential count) below 4 × 109/L (4000/μL), absence of significant lymphadenopathy (lymph nodes must be < 1.5 cm), absence of splenomegaly and hepatomegaly, absence of constitutional symptoms, normal blood counts, and bone marrow sample must be at least normocellular for age, with less than 30% of nucleated cells being lymphocytes. Lymphoid nodules should be absent.
Time Frame: 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Chemotherapy
Number analyzed (Participants) | 22
percentage of patients | 36

ADVERSE EVENTS:
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=22)
Fatal septic shock secondary to bacteremia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=22)
grade 3/4 neutropenia (Blood and lymphatic system disorders) | 13 — grade 3/4 neutropenia during FR: 59% and during lenalidomide: 27%
grade 1/2 anemia (Blood and lymphatic system disorders) | 12 — grade 1/2 anemia during FR: 54% ; and during lenalidomide: 20%
grade 3/4 anemia (Blood and lymphatic system disorders) | 4 — grade 3/4 anemia during FR: 18% and during lenalidomide: 0%
grade 1/2 neutropenia (Blood and lymphatic system disorders) | 2 — grade 1/2 neutropenia during FR: 9% and during lenalidomide: 27%
grade 1/2 thrombocytopenia (Blood and lymphatic system disorders) | 2 — grade 1/2 thrombocytopenia during FR: 9% and during lenalidomide: 40%
grade 3/4 thrombocytopneia (Blood and lymphatic system disorders) | 4 — grade 3/4 thrombocytopenia during FR: 18% and during lenalidomide: 0%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No